CLINICAL TRIAL: NCT00383253
Title: A Randomized, Open-Label, Parallel Group, Fixed Energy Deficit Methodology Trial to Characterize Early Efficacy Biomarkers During Treatment of Obesity in Adult, Obese, Male Subjects.
Brief Title: Methods Study to Characterize Early Indicators of Weight Loss in People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: University of Adelaide (Other); Royal Adelaide Hospital (Other)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A9001342
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2009-03-23 (Estimated); Status verified 2009-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 10% (Experimental)
  Interventions: Behavioral: caloric restriction - 10%
- 25% (Experimental)
  Interventions: Behavioral: caloric restriction - 25%
- 50% (Experimental)
  Interventions: Behavioral: caloric restriction - 50%
- Control (Placebo Comparator)
  Interventions: Behavioral: caloric restriction - Control

INTERVENTIONS:
Behavioral: caloric restriction - 10% — Subjects maintained on 10% caloric restriction (caloric intake = 90% of baseline)
  Arms: 10%
Behavioral: caloric restriction - 25% — Subjects maintained on 25% caloric restriction (caloric intake = 75% of baseline)
  Arms: 25%
Behavioral: caloric restriction - 50% — Subjects maintained on 50% caloric restriction (caloric intake = 50% of baseline)
  Arms: 50%
Behavioral: caloric restriction - Control — Subjects maintained on their baseline caloric intake (caloric restriction = none)
  Arms: Control

SUMMARY:
Methods study to characterize early indicators of weight loss in people.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >=18 years of age with BMI >= 30 and < 40 kg/m2

Exclusion Criteria:

* Females, those with illnesses expected to cause weight loss, those without stable body weight within 3 months of screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2006-10; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of varying degrees of controlled, 1-month, caloric restriction on weight loss, and response of known circulating, candidate biomarkers | Throughout trial

SECONDARY OUTCOMES:
To evaluate the time course, magnitude and biomarkers of metabolic compensation as well as assessment of well being (via questionnaires) following varying degrees of controlled, 1-month, caloric restriction | Throughout trial

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Australia (2):
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, North Adelaide, South Australia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001342&StudyName=Methods%20study%20to%20characterize%20early%20indicators%20of%20weight%20loss%20in%20people.